CLINICAL TRIAL: NCT03527537
Title: Gestational Diabetes and Pharmacotherapy (GAP) - A Randomized Controlled Trial Investigating Timing of Pharmacotherapy Initiation for Patients With Gestational Diabetes
Brief Title: Gestational Diabetes and Pharmacotherapy (GAP)
Acronym: GAP
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Anna Palatnik, MD, Assistant Professor, Medical College of Wisconsin
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRO00030802
Record Dates: First submitted 2018-04-24; First posted 2018-05-17 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Gestational Diabetes
MeSH Terms: conditions — Diabetes, Gestational | interventions — Insulin

STUDY DESIGN:
Intervention Model Description: This will be a randomized, controlled trial of 284 women with a diagnosis of GDM. Women will be consented and randomized at the time of their diagnosis. All women with GDM will receive counseling regarding diet and exercise and instructions on self-monitoring blood glucose values. The investigators will apply cutoffs of 95 mg/dL for fasting and 120 mg/dL for 2-hour post-prandial levels. Once randomized, the first treatment arm will be assigned to a limit of 20% abnormal values before we start treatment and to titrate up dosages as needed, while using the 20% threshold of abnormal CBG values at each subsequent review of glucose log. To specify, if more than 20% of values for the week are elevated, treatment would be initiated. Once treatment is initiated, the dosage of medication will be adjusted with cutoff of 20% of abnormal values per week. The second treatment arm will utilize the same protocol, however, the limit to start medications or adjust dosages will be 40% abnormal values.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- 20% cutoff group (Active Comparator): Treatment intervention will be initiated with insulin if 20% cutoff of abnormal values is reached. Medication dosages will depend on the physician's discretion.
  Interventions: Drug: Insulin
- 40% cutoff group (Active Comparator): Treatment intervention will be initiated with insulin if 40% cutoff of abnormal values is reached. Medication dosages will depend on the physician's discretion.
  Interventions: Drug: Insulin

INTERVENTIONS:
Drug: Insulin — Insulin may be administered base on glucose log values. The dosing of the insulin will be determined by the provider using typical management of gestational diabetes.

SUMMARY:
The goal of this study is to compare two different thresholds for initiation of medical treatment for GDM. Pregnant women diagnosed with GDM will be randomized to either start pharmacotherapy when they have reached at least 20% or at least 40% of capillary blood glucose (CBG) values above the target goal. The investigators hypothesize that a lower threshold of 20% elevated CBG levels, compared to 40%, will lead to lower rates of obstetric and medical complications.

DETAILED DESCRIPTION:
Gestational diabetes mellitus (GDM) affects 5-8% of pregnant women, many of whom will require treatment beyond diet and exercise. Despite this high prevalence, there is no consensus regarding the glycemic threshold for conversion from diet to medical treatment for GDM. No randomized studies have been performed on how to define failure with diet and exercise and currently, the need to start insulin or oral hypoglycemic agents is at the provider's discretion. It is important to establish criterion of pharmacotherapy initiation for GDM in pregnancy as GDM under-treatment leads to increased rates of adverse obstetric outcomes associated with poor glycemic control including macrosomia, pre-eclampsia, cesarean delivery, shoulder dystocia, birth trauma, neonatal hypoglycemia and hyperbilirubinemia, childhood obesity and metabolic syndrome in the offspring. In contrast, overtreatment for women comes at increased cost due to overutilization of resources, increased expense, and adverse effects of the medications themselves.

The goal of this study is to compare two different thresholds for initiation of medical treatment for GDM. Pregnant women diagnosed with GDM (N=416) will be randomized to either start pharmacotherapy when they have reached at least 20% or at least 40% of capillary blood glucose (CBG) values above the target goal. The investigators hypothesize that a lower threshold of 20% elevated CBG levels, compared to 40%, will lead to lower rates of obstetric and medical complications.

Aim 1: Determine the effect of earlier insulin initiation (20% threshold) for GDM management on adverse neonatal and maternal outcomes associated with GDM.

Hypothesis 1.1: The composite adverse neonatal outcome associated with GDM (LGA, macrosomia, birth trauma, preterm birth, neonatal hypoglycemia, and hyperbilirubinemia) will be lower in earlier insulin initiation compared with the active control group.

Hypothesis 1.2: Preeclampsia and cesarean birth frequencies will be lower in earlier insulin initiation compared with the active control group.

Hypothesis 1.3: The composite neonatal and maternal outcomes will not differ between racial and ethnic groups within each study group.

Aim 2:Assess the safety of earlier insulin initiation in pregnant patients and their neonates.

Hypothesis 2.1: The SGA rate will be higher in earlier insulin initiation compared with the active control group; however, in both groups it will be lower than the national rate of 10%. Hypothesis 2.2: Maternal hypoglycemia and perinatal death will not differ between groups.

Aim 3:Determine the effect of earlier insulin initiation on patient-reported outcomes using standardized measures and qualitative interviews.

Hypothesis 3: Anxiety, depression, perceived stress and diabetes self-efficacy will be better in patients randomized to earlier insulin initiation compared with the active control group.

ELIGIBILITY:
Inclusion Criteria:

* Viable singleton pregnancy
* Age >= 18 years old
* Diagnosed with gestational diabetes mellitus
* Able to communicate in English

Exclusion Criteria:

* Pre-gestational diabetes
* Significantly abnormal GDM testing, suggestive of the presence of pre-gestational diabetes, either with fasting values >=126 mg/dL or 2-hour post-prandial levels >=200 mg/dL
* Patients who check blood sugars on average less than 2 times per day after appropriate counseling
* Already started pharmacotherapy prior to referral to the study

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Only women will be randomized as this is a pregnancy-focused study
Enrollment: 416 (Estimated)
Dates: Start 2021-05-04 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Composite Neonatal Outcome | The data will be collected up to 6 weeks of life
  Our primary outcome will be a composite adverse neonatal outcome associated with gestational diabetes:
  large-for-gestational age macrosomia birth trauma preterm birth neonatal hypoglycemia hyperbilirubinemia

SECONDARY OUTCOMES:
Cesarean Delivery Rate | The data will be collected up to 6 weeks postpartum
  Our secondary outcome will be to compare the rates of cesarean delivery between two thresholds for medical treatment initiation for GDM.
Preeclampsia | The data will be collected up to 6 weeks postpartum

CONTACTS AND LOCATIONS:
Locations (1):
- Medical College of Wisconsin, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] ACOG Practice Bulletin No. 190: Gestational Diabetes Mellitus. Obstet Gynecol. 2018 Feb;131(2):e49-e64. doi: 10.1097/AOG.0000000000002501. PMID 29370047
- [Background] Hartling L, Dryden DM, Guthrie A, Muise M, Vandermeer B, Donovan L. Benefits and harms of treating gestational diabetes mellitus: a systematic review and meta-analysis for the U.S. Preventive Services Task Force and the National Institutes of Health Office of Medical Applications of Research. Ann Intern Med. 2013 Jul 16;159(2):123-9. doi: 10.7326/0003-4819-159-2-201307160-00661. PMID 23712381
- [Background] Langer O, Yogev Y, Most O, Xenakis EM. Gestational diabetes: the consequences of not treating. Am J Obstet Gynecol. 2005 Apr;192(4):989-97. doi: 10.1016/j.ajog.2004.11.039. PMID 15846171
- [Background] Crowther CA, Hiller JE, Moss JR, McPhee AJ, Jeffries WS, Robinson JS; Australian Carbohydrate Intolerance Study in Pregnant Women (ACHOIS) Trial Group. Effect of treatment of gestational diabetes mellitus on pregnancy outcomes. N Engl J Med. 2005 Jun 16;352(24):2477-86. doi: 10.1056/NEJMoa042973. Epub 2005 Jun 12. PMID 15951574
- [Background] Landon MB, Spong CY, Thom E, Carpenter MW, Ramin SM, Casey B, Wapner RJ, Varner MW, Rouse DJ, Thorp JM Jr, Sciscione A, Catalano P, Harper M, Saade G, Lain KY, Sorokin Y, Peaceman AM, Tolosa JE, Anderson GB; Eunice Kennedy Shriver National Institute of Child Health and Human Development Maternal-Fetal Medicine Units Network. A multicenter, randomized trial of treatment for mild gestational diabetes. N Engl J Med. 2009 Oct 1;361(14):1339-48. doi: 10.1056/NEJMoa0902430. PMID 19797280
- [Background] Athukorala C, Crowther CA, Willson K; Austrailian Carbohydrate Intolerance Study in Pregnant Women (ACHOIS) Trial Group. Women with gestational diabetes mellitus in the ACHOIS trial: risk factors for shoulder dystocia. Aust N Z J Obstet Gynaecol. 2007 Feb;47(1):37-41. doi: 10.1111/j.1479-828X.2006.00676.x. PMID 17261098
- [Background] Gilbert WM, Nesbitt TS, Danielsen B. Associated factors in 1611 cases of brachial plexus injury. Obstet Gynecol. 1999 Apr;93(4):536-40. doi: 10.1016/s0029-7844(98)00484-0. PMID 10214829
- [Background] Boney CM, Verma A, Tucker R, Vohr BR. Metabolic syndrome in childhood: association with birth weight, maternal obesity, and gestational diabetes mellitus. Pediatrics. 2005 Mar;115(3):e290-6. doi: 10.1542/peds.2004-1808. PMID 15741354
- [Background] Clausen TD, Mathiesen ER, Hansen T, Pedersen O, Jensen DM, Lauenborg J, Schmidt L, Damm P. Overweight and the metabolic syndrome in adult offspring of women with diet-treated gestational diabetes mellitus or type 1 diabetes. J Clin Endocrinol Metab. 2009 Jul;94(7):2464-70. doi: 10.1210/jc.2009-0305. Epub 2009 May 5. PMID 19417040
- [Background] Dabelea D, Snell-Bergeon JK, Hartsfield CL, Bischoff KJ, Hamman RF, McDuffie RS; Kaiser Permanente of Colorado GDM Screening Program. Increasing prevalence of gestational diabetes mellitus (GDM) over time and by birth cohort: Kaiser Permanente of Colorado GDM Screening Program. Diabetes Care. 2005 Mar;28(3):579-84. doi: 10.2337/diacare.28.3.579. PMID 15735191
- [Background] American Diabetes Association. Diagnosis and classification of diabetes mellitus. Diabetes Care. 2012 Jan;35 Suppl 1(Suppl 1):S64-71. doi: 10.2337/dc12-s064. No abstract available. PMID 22187472
- [Background] HAPO Study Cooperative Research Group; Metzger BE, Lowe LP, Dyer AR, Trimble ER, Chaovarindr U, Coustan DR, Hadden DR, McCance DR, Hod M, McIntyre HD, Oats JJ, Persson B, Rogers MS, Sacks DA. Hyperglycemia and adverse pregnancy outcomes. N Engl J Med. 2008 May 8;358(19):1991-2002. doi: 10.1056/NEJMoa0707943. PMID 18463375
- [Background] Kim C, Newton KM, Knopp RH. Gestational diabetes and the incidence of type 2 diabetes: a systematic review. Diabetes Care. 2002 Oct;25(10):1862-8. doi: 10.2337/diacare.25.10.1862. PMID 12351492
- [Background] Caissutti C, Berghella V. Scientific Evidence for Different Options for GDM Screening and Management: Controversies and Review of the Literature. Biomed Res Int. 2017;2017:2746471. doi: 10.1155/2017/2746471. Epub 2017 Apr 10. PMID 28497042
- [Background] Rumbold AR, Crowther CA. Guideline use for gestational diabetes mellitus and current screening, diagnostic and management practices in Australian hospitals. Aust N Z J Obstet Gynaecol. 2001 Feb;41(1):86-90. doi: 10.1111/j.1479-828x.2001.tb01301.x. PMID 11284655
- [Background] American Diabetes Association. 13. Management of Diabetes in Pregnancy. Diabetes Care. 2017 Jan;40(Suppl 1):S114-S119. doi: 10.2337/dc17-S016. No abstract available. PMID 27979900